CLINICAL TRIAL: NCT02768870
Title: Mitral TRans-Apical neoChordal Echo-guided Repair (TRACER) Trial
Brief Title: CE Mark Study for the Harpoon Medical Device
Acronym: TRACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMCE-1002-00k
Record Dates: First submitted 2016-04-20; First posted 2016-05-11 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Mitral Valve Regurgitation; Mitral Valve Prolapse; Mitral Valve Insufficiency
Keywords: Mitral Valve Repair; Transapical; Artificial Chordae
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Harpoon Medical Device (Experimental): This is a prospective, single arm, nonrandomised, multi-center EU study to demonstrate the performance and safety of the Harpoon Medical device in patients with degenerative MR.
  Interventions: Device: Harpoon Artificial ePTFE Chords

INTERVENTIONS:
Device: Harpoon Artificial ePTFE Chords — It is anticipated that use of the Harpoon device could achieve similar outcomes to open cardiac surgery while decreasing the invasiveness of mitral valve repair.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Harpoon Medical device. It is anticipated, that the Harpoon Medical device will provide advantages over current surgical interventions including: 1) a small minimally invasive incision, 2) no sternotomy, 3) no cardiopulmonary bypass, 4) no aortic manipulation, 5) a direct path to the valve plane, 6) performed on a beating heart, 7) real-time TOE-guided chordal length adjustment and 8) less complicated procedure that is teachable and adoptable.

DETAILED DESCRIPTION:
The device is designed to reduce the degree of mitral regurgitation by delivering and anchoring artificial chordae tendineae to the affected mitral valve leaflet(s) in a beating heart.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient referred for mitral valve surgery
* Presence of severe MR as read on an echocardiographic study performed within 60 days prior to procedure
* Estimated post-ePTFE chordae tendineae implantation coaptation surface is adequate in the judgment of the operating surgeon and the patient eligibility committee
* Degenerative mitral valve disease
* Patient is able to sign informed consent and able to return for follow-up and is capable of participating in all testing associated with this clinical investigation
* Women of child-bearing potential have a negative pregnancy test

Exclusion Criteria:

* Age < 18 years
* Infective endocarditis
* Anterior or bileaflet prolapse
* Functional MR
* History of Mediastinal Radiation
* Inflammatory (rheumatic) valve disease
* Requirement for concomitant cardiac surgery (e.g., coronary artery bypass grafting (CABG), aortic valve surgery, etc.)
* Symptomatic coronary artery disease
* Cardiogenic shock at the time of enrollment
* ST segment elevation myocardial infarction requiring intervention within 30 days prior to enrollment
* Evidence of cirrhosis or hepatic synthetic failure
* Pregnancy at the time of enrollment (women of child bearing age should have negative pregnancy within 14 days of surgery)
* Severe pulmonary hypertension (PA systolic pressure > 70 mmHg)
* Previous cardiac surgery, or surgery on the left pleural space
* Left ventricular, atrial or appendage thrombus
* Severely calcified mitral leaflets
* Recent stroke (< 6 months) with permanent impairment
* EuroScore (for mitral valve repair) > 8%
* Patients with contraindications to Transoesophageal echocardiography
* Severe left or right ventricular dysfunction
* NYHA Class IV
* Renal insufficiency CKD stage 3b or worse (GFR < 45 ml/min/1.73 m2)
* Patient is participating in another clinical study for which follow-up is currently ongoing. (Co-enrollment in an investigational device or interventional study)
* Patient with non-cardiac co-morbidities and life expectancy < 1 year
* Patient has a condition or conditions that, in the opinion of the Investigator, preclude participation, including willingness to comply with all follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino Gerosa, MD, Principal Investigator — University Hospital Padova; Ottavio Alfieri, MD, Principal Investigator — OSR San Raffaele Hospital; Alison Duncan, MD, Principal Investigator — The Royal Brompton Hospital
Locations (4):
- Italy (2):
  - Ospedale San Raffaele Hospital, Milan
  - University Hospital Padova, Padua
- United Kingdom (2):
  - The Royal Brompton and Harefield NHS Foundation Trust, London
  - University Hospital Southampton NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Result] Gammie JS, Bartus K, Gackowski A, D'Ambra MN, Szymanski P, Bilewska A, Kusmierczyk M, Kapelak B, Rzucidlo-Resil J, Moat N, Duncan A, Yadev R, Livesey S, Diprose P, Gerosa G, D'Onofrio A, Pitterello D, Denti P, La Canna G, De Bonis M, Alfieri O, Hung J, Kolsut P. Beating-Heart Mitral Valve Repair Using a Novel ePTFE Cordal Implantation Device: A Prospective Trial. J Am Coll Cardiol. 2018 Jan 2;71(1):25-36. doi: 10.1016/j.jacc.2017.10.062. Epub 2017 Nov 1. PMID 29102688
- [Derived] Gammie JS, Bartus K, Gackowski A, Szymanski P, Bilewska A, Kusmierczyk M, Kapelak B, Rzucidlo-Resil J, Duncan A, Yadav R, Livesey S, Diprose P, Gerosa G, D'Onofrio A, Pittarello D, Denti P, La Canna G, De Bonis M, Alfieri O, Hung J, Kolsut P, D'Ambra MN. Safety and performance of a novel transventricular beating heart mitral valve repair system: 1-year outcomes. Eur J Cardiothorac Surg. 2021 Jan 4;59(1):199-206. doi: 10.1093/ejcts/ezaa256. PMID 33038223

RESULTS

PARTICIPANT FLOW:
Groups:
- Harpoon Medical Device: Safety and Performance study of the Harpoon Medical Device in subjects with degenerative mitral regurgitation.
Period: Overall Study
Arm/Group | Harpoon Medical Device
Started (Enrolled in Study) | 26
Implanted With Device | 24
Discharge | 26
30 Days | 26
6 Months | 25
12 Months | 23
18 Months | 23
24 Months | 21
30 Months | 19
36 Months | 17
48 Months | 15
60 Months | 14
Completed | 14
Not Completed | 12
Not completed — Death | 1
Not completed — Reoperation | 6
Not completed — Lost to Follow-up | 1
Not completed — Exit | 4

BASELINE CHARACTERISTICS:
Population: Subjects enrolled in the trial.
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject's Procedural Success During the First 30 Days
Description: Procedural success was defined as the patient leaving the operating room with a successful implant of one or more ePTFE cords on the mitral valve and reduced mitral regurgitation from severe to </=moderate at the conclusion of the procedure and at 30 days post-procedure.
Time Frame: End of procedure through 30 days
Population: This outcome is reported for enrolled subjects where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Participants | 23

2. Primary Outcome: Percentage of Subject's With Freedom From Serious Adverse Events (SAE) </= 30 Days
Description: Subject's freedom from Serious Adverse Events during the ePTFE implantation procedure and at 30 days follow-up. Time to events were estimated by Kaplan-Meier method.
Time Frame: Procedure and 30 days
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
percentage of subjects
  KM estimate: Procedure | 92.3 [82.1 to 100.0]
  KM estimate: 30 Days | 57.7 [38.7 to 76.7]

3. Primary Outcome: Subject's Serious Adverse Events (SAE) Through Discharge
Description: Number of Participants experiencing a Serious Adverse Event (SAE) through time of Discharge.
Time Frame: Discharge, an average of 5 days post implant
Population: This outcome is reported for enrolled subjects where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Participants | 6

4. Secondary Outcome: Subject's Severity of Mitral Regurgitation Over Time
Description: Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation. The numbers on the scale are reflected as follows: 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak.
  Higher numbers on the scale show a worsening outcome.
Time Frame: 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
Population: This outcome is reported for subjects who received the Harpoon Medical Device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 24
Participants
  6 month follow-up: number analyzed (Participants) | 23
  6 month follow-up: None | 9
  6 month follow-up: Trace | 3
  6 month follow-up: Mild | 6
  6 month follow-up: Moderate | 2
  6 month follow-up: Severe | 3
  12 month follow-up: number analyzed (Participants) | 20
  12 month follow-up: None | 3
  12 month follow-up: Trace | 6
  12 month follow-up: Mild | 6
  12 month follow-up: Moderate | 4
  12 month follow-up: Severe | 1
  18 month follow-up: number analyzed (Participants) | 7
  18 month follow-up: None | 2
  18 month follow-up: Trace | 4
  18 month follow-up: Mild | 0
  18 month follow-up: Moderate | 1
  18 month follow-up: Severe | 0
  24 month follow-up: number analyzed (Participants) | 19
  24 month follow-up: None | 1
  24 month follow-up: Trace | 9
  24 month follow-up: Mild | 3
  24 month follow-up: Moderate | 3
  24 month follow-up: Severe | 3
  30 month follow-up: number analyzed (Participants) | 14
  30 month follow-up: None | 4
  30 month follow-up: Trace | 4
  30 month follow-up: Mild | 0
  30 month follow-up: Moderate | 2
  30 month follow-up: Severe | 4
  36 month follow-up: number analyzed (Participants) | 11
  36 month follow-up: None | 1
  36 month follow-up: Trace | 4
  36 month follow-up: Mild | 3
  36 month follow-up: Moderate | 1
  36 month follow-up: Severe | 2

5. Secondary Outcome: Percentage of Subject's With Freedom From Serious Adverse Events (SAE) Post-implant > 30 Days
Description: Subject's freedom from Serious Adverse Events at >30 days post-implant. Time to events were estimated by Kaplan-Meier method.
Time Frame: 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
percentage of subjects
  KM estimate: 6 months | 46.2 [27.0 to 65.3]
  KM estimate:12 months | 38.5 [19.8 to 57.2]
  KM estimate:18 months | 38.5 [19.8 to 57.2]
  KM estimate:24 months | 38.5 [19.8 to 57.2]
  KM estimate:30 months | 38.5 [19.8 to 57.2]
  KM estimate:36 months | 38.5 [19.8 to 57.2]

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through 60 months post implant.
Groups:
- Harpoon Medical Device: Safety and Performance study of the enrolled cohort of the Harpoon clinical trial.
Arm/Group | Harpoon Medical Device
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 19/26
Other Adverse Events (participants affected / at risk) | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harpoon Medical Device (N=26)
Arrhythmia - Persistent atrial fibrillation (Cardiac disorders) | 8 (8)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 6 (6)
ePTFE cordal rupture (Product Issues) | 5 (5)
Blood sepsis (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular - Other (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (2)
Pleural effusion - Left (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Regurgitation - Mitral-indeterminate +4 (Cardiac disorders) | 1 (1)
DAMAGE TO THE NATIVE MITRAL VALVE APPARATUS CHORD (Product Issues) | 2 (2)
BLEEDING - NEUROLOGICAL - MINOR (E.G. CVA) (Blood and lymphatic system disorders) | 1 (1)
REGURGITATION - MITRAL-INDETERMINATE +2 (Cardiac disorders) | 1 (1)
CANCER - NEWLY DIAGNOSED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MUSCULAR SKELETAL/DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 1 (1)
BLEEDING - CARDIOVASCULAR - MAJOR (Blood and lymphatic system disorders) | 1 (1)
ARRHYTHMIA - ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
PERFORATION, TEAR OR INJURY - VENTRICULAR MAJOR (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harpoon Medical Device (N=26)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 7 (12)
Arrhythmia - AV block - 1st degree (Cardiac disorders) | 3 (3)
Genitourinary - Other (Renal and urinary disorders) | 2 (2)
MUSCULAR SKELETAL/DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 2 (3)
BLOOD/LYMPHATIC - OTHER (Blood and lymphatic system disorders) | 2 (2)
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 1 (1)
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 2 (2)
ARRHYTHMIA - AV BLOCK - 3RD DEGREE (Cardiac disorders) | 1 (1)
ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT (Cardiac disorders) | 1 (1)
ARRHYTHMIA - TACHYCARDIA - VENTRICULAR (Cardiac disorders) | 1 (1)
REGURGITATION - MITRAL-INDETERMINATE +1 (Cardiac disorders) | 1 (1)
REGURGITATION - MITRAL-INDETERMINATE +2 (Cardiac disorders) | 1 (1)
REGURGITATION - MITRAL-INDETERMINATE +3 (Cardiac disorders) | 1 (1)
REGURGITATION - MITRAL-INDETERMINATE +4 (Cardiac disorders) | 1 (1)
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 1 (1)
INFECTION/INFLAMMATION - OTHER (Infections and infestations) | 1 (1)
METABOLIC COMPLICATIONS (Metabolism and nutrition disorders) | 1 (1)
STERNAL WOUND/THORACIC INFECTION (Infections and infestations) | 1 (1)
WOUND INFECTION - OTHER (Infections and infestations) | 1 (1)
PLEURAL EFFUSION - LEFT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE - PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish site data until first multi-center publication. Publications will be submitted to Sponsor for review 60 days prior to publication/dissemination. Sponsor may ask for a 6-month delay of publication to protect proprietary information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02768870/Prot_SAP_001.pdf